CLINICAL TRIAL: NCT04586530
Title: Mobile Device CBT for Chemotherapy-Related Cognitive Dysfunction: A Multi-Center Randomized Controlled Trial
Brief Title: Telehealth and Memory Study
Acronym: TAMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Donna Posluszny, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCC 20-064; R01CA244673-01A1 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-related Cognitive Dysfunction
Keywords: Memory and Attention Adaptation Training (MAAT); cognitive-impairment; cancer survivorship
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment; Cognition Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memory and Attention Adaptation Training (MAAT) (Experimental): A videoconference-delivered cognitive-behavioral therapy (CBT) for treatment of chemotherapy-related cognitive dysfunction (CRCD) among cancer survivors consisting of 8 weekly 45-minute visits with a survivor workbook, that targets: 1) enhancement of survivor self-awareness of "at risk" situations where memory failures occur; 2) emotion regulation through modification of survivor causal attributions and negative cognitive appraisals of memory failures; and 3) training in compensatory strategies to improve performance on daily tasks for which memory.
  Interventions: Behavioral: Memory and Attention Adaptation Training (MAAT)
- Supportive Therapy (ST) (Active Comparator): Standard attention control condition therapy for treatment of chemotherapy-related cognitive dysfunction (CRCD) among cancer survivors consisting of 8, 45-minutes visits. ST, emphasizes "non-specific" psychotherapeutic factors of clinician-participant alliance: empathy, support and warmth. ST will be directed at concerns with cancer survivorship and CRCD. Clinicians will set expectations with ST participants that they will be provided validation of experience, support, and encouragement of building their own coping resources if asked directly about what to do about cognitive problems. ST emphasizes reflective listening to help deepen knowledge of the emotional experience of the participant.
  Interventions: Behavioral: Supportive Therapy (ST)

INTERVENTIONS:
Behavioral: Memory and Attention Adaptation Training (MAAT) — A cognitive-behavioral therapy (CBT) for treatment of chemotherapy-related cognitive dysfunction (CRCD) among cancer survivors.
  Arms: Memory and Attention Adaptation Training (MAAT)
Behavioral: Supportive Therapy (ST) — Standard attention control condition therapy for treatment of chemotherapy-related cognitive dysfunction (CRCD) among cancer survivors.
  Arms: Supportive Therapy (ST)

SUMMARY:
The overall purpose of this trial is to confirm the efficacy of Memory and Attention Adaptation Training (MAAT), a cognitive-behavioral therapy (CBT) for treatment of chemotherapy-related cognitive dysfunction among (female or male) breast cancer survivors. This is a multi-center, multi-clinician randomized control trial (MAAT vs. supportive therapy attention control condition). This trial will also evaluate a sub-sample of survivors pre-and post treatment with functional magnetic resonance imaging (fMRI) in a working memory task to evaluate pre-to-post treatment brain activation patterns to elucidate underlying mechanisms of clinical therapeutic change.

DETAILED DESCRIPTION:
The primary aim of this multi-site, multi-clinician randomized controlled trial is to determine if Memory and Attention Adaptation Training (MAAT), a cognitive-behavioral therapy (CBT) intervention, can improve self-reported and objectively measured cognitive functioning in breast cancer survivors who previously received chemotherapy. Breast cancer survivors (Stage I-III) who were treated with chemotherapy 1-5 years prior to enrollment and who have subjective cognitive complaints may be eligible for this study. After eligibility is confirmed, participants will complete baseline assessments of subjective and objective memory and attention functioning as well as behavioral rating scales, and will be randomized to MAAT or Supportive Therapy (ST; to control for therapist time and attention) for 8 weeks. Both treatments (MAAT and ST) will be delivered through videoconferencing using mobile (smartphone, laptop or other electronic device) in order to reduce survivor travel or time away from work or family. Data collection methods will include telephone- and web-administered measures of subjective and objective cognitive function, as well as various behavioral ratings. Outcome assessments will be conducted post-treatment and at 6-month follow-up. It is hypothesized that MAAT participants will have significantly improved scores of self-reported cognitive impairments and objective neurocognitive test scores (on verbal memory and processing speed) at post-treatment and 6-month follow-up compared to participants randomized to ST. In addition, willing and eligible participants will be asked to complete a functional MRI working memory task at baseline and post-treatment, to examine whether those who receive MAAT show greater increase in brain network activation than those who receive ST. This may advance understanding of the neural mechanisms underlying improvement of objective and self-reported cognitive function after chemotherapy. The sample size (n=100/group) will allow for a 10-15% drop out-rate and still provide 80% power to detect group differences using two (Group: MAAT vs. ST) by 3 (time: baseline, posttreatment, 6-month follow-up) ANCOVA at alpha=0.05. Potential baseline differences between MAAT and ST groups on primary outcome variables or other factors that may affect cognition (e.g., anxiety, fatigue or depression) will be evaluated as potential covariates, although such differences due to randomization are not anticipated.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stage I-III breast cancer
2. 1-5 years post-treatment and currently disease free
3. Treatment involved adjuvant or neoadjuvant chemotherapy
4. Report cognitive problems of memory and concentration attributed to chemotherapy with a score of 10 or below on the FACT-Cog Impact on Quality of Life Scale (a score ~1SD below pre-chemotherapy treatment norms; this criterion was used in our prior R21 study, ensures a clinically meaningful level of cognitive concerns,41 and discriminates high and low PCI scores in prior research42)
5. Able to speak and read English
6. Age >18
7. Able to provide IRB-approved written informed consent
8. Willing to use videoconferencing.

Exclusion Criteria:

1. Previous CNS radiation, intrathecal therapy, or CNS-involved surgery
2. Previous cancer history with the exception of non-melanoma skin cancer
3. Previous exposure to chemotherapy with another cancer or due to other medical condition (e.g., methotrexate exposure for treatment of rheumatoid arthritis)
4. Significant neurodevelopmental, neurobehavioral, or medical risk factors likely to affect cognitive functioning (e.g., history of neurological disorder or TBI of greater than mild severity, such as loss of consciousness >30 minutes, medical disorder that is unstable or likely to affect cognition such as metabolic disorder, heart attack or stroke, uncontrolled diabetes or endocrine dysfunction)
5. Currently meeting DSM-5 mental disorder criteria, including but not limited to neurodevelopmental, substance abuse, mood (e.g., Maj.Dep), anxiety, or psychotic disorders
6. Scoring 3 or below on the 6-item cognitive screen designed to detect severe memory disorders;43
7. Severe uncorrected sensory impairment (severe hearing or visual impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
FACT-Cog PCI | At Baseline, Post-Treatment (8 weeks) and 6-Month Follow-up
  The FACT-Cog is a 37-item self-report measure that uses 5- point (0-4) Likert-type ratings that produce four scales: 1) Impact on quality of life; 2) Perceived cognitive impairments; 3) Comments from others; and 3) Perceived cognitive abilities. Higher scores indicate better function and quality of life on each scale. While each scale is scored and interpreted separately, they comprise the total Fact-cog assessment. The FACT-Cog has good evidence of reliability and construct validity. We are assessing change in PCI -- from baseline to post-treatment, to 6-month follow-up-- as our primary measure of outcome.

SECONDARY OUTCOMES:
California Verbal Learning Test-3 (CVLT-3) | At Baseline, Post-Treatment (8 weeks) and 6-Month Follow-up
  The California Verbal Learning Test is a neuropsychological assessment of episodic verbal and working memory and processing speed. Participants listen to series of words and is then asked to recall the terms and the category to which they belong. This assessment attempts to measure how much a subject learned and also reveal strategies employed and the types of errors made. Higher CVLT-3 scores are associated with better memory and processing function.
Controlled Oral Word Association Test (COWAT) | At Baseline, Post-Treatment (8 weeks) and 6-Month Follow-up
  The Controlled Oral Word Association Test (COWAT), is a neuropsychological measure of verbal fluency. The COWAT consists of three word conditions. Participants are asked to produce as many words as they can that begin with the F, A, or S within a 1 minute time period. The total number of words that the individual is able to produce provides a score. Typically, if someone scores less than 17 words, the test administrator will use additional tests to further evaluate cognition.
Digit Span test | At Baseline, Post-Treatment (8 weeks) and 6-Month Follow-up
  The Digit Span test is a neurocognitive subset of both the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Memory Scales (WMS) that assesses working memory. Participants read a sequence of numbers and are asked to repeat the same sequence back to the examiner in order (forward span) or in reverse order (backward span). This assessment generates three "raw" scores and one overall age-appropriate normed (standard) score. Higher scores indicate better working memory and neurocognitive function.
Symbol Digit Modalities Test (SDMT) | At Baseline, Post-Treatment (8 weeks) and 6-Month Follow-up
  The Symbol Digit Modalities Test (SDMT) is a neurocognitive screening instrument used to assess neurological dysfunction. Participants are required to use a coded key to match nine abstract symbols paired with numerical digits. Ten (10) practice items before commencing the test. The final score is the correct number of substitutions in 90 seconds, and scores range between 0 and 110. Higher scores indicate better neurocognitive functioning.
functional Magnetic Resonance Imaging (fMRI) | At Baseline and Post-Treatment (8 weeks)
  fMRI assessment of a working memory task (N-Back) will assess brain activation patterns through detection in bloodflow changes. The fMRI N-Back working memory task has been demonstrated to reflect increased activation in response to MAAT treatment among individuals with traumatic brain injury.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Ferguson, PhD, Principal Investigator — St. Jude Children's Research Hospital; Donna Posluszny, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NIH funded study - public database
Supporting Information: Study Protocol, SAP
Time Frame: We anticipate a completed data set in approximately December of 2025 and will make de-identified data available to qualified investigators for a period of 3 years after publication of primary results in a peer reviewed journal.
Access Criteria: De-identified data sharing criteria include (for quality assurance): 1) Qualified researchers who have obtained IRB approval from their institution; 2) Sign a Data Use Agreement (DUA); 3) Agree to NIH, IRB policies and HIPAA requirements regarding privacy, data security and ethical practices; 4) The DUAs will ensure that data will be used only for the specific research purposes outlined in the DUA; 5) No personally identifiable or protected health information will be shared outside of University of Pittsburgh/Indiana University research staff who have a need to know this information for the purposes of the study; 6) Individual participant's data will not be disseminated; 7) Data access will be protected under security measures including encryption and password protection, and that the data will be destroyed or returned to the University of Pittsburgh/Indiana University study team after completion of relevant analyses. Collaborative analyses with project investigators are encouraged.

DOCUMENTS (1):
  • Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT04586530/ICF_000.pdf